CLINICAL TRIAL: NCT06164613
Title: Use of Cinnamomum Verum Extract Versus Placebo for Induction of Labor and Reduction of Physiological Phase 2-3 of Labor. Double-blind Randomized Clinical Trial. CINNALAB TRIAL
Brief Title: Use of Cinnamomum Verum for Induction of Labor. Double Blind Randomized Clinical Trial
Acronym: CINNALAB
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Universidad Nacional Autonoma de Honduras (Other)
Responsible Party: Principal Investigator, Ricardo A Gutierrez Ramirez, MD, MSc, FACOG, Professor, research coordinator of the postgraduate course in gynecology and obstetrics, Universidad Nacional Autonoma de Honduras
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: CV-LT-01-2023
Record Dates: First submitted 2023-12-01; First posted 2023-12-11 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Labor Onset and Length Abnormalities; First Birth
Keywords: cinnamon oil, bark; labor onset; nulliparity
MeSH Terms: interventions — Rapeseed Oil

STUDY DESIGN:
Intervention Model Description: parallel group, efficacy, randomized, placebo-controlled, double-blind clinical trial.
Who Masked: Participant, Care Provider, Investigator
Masking Description: The masking of the treatment will be carried out by a person external to the study; in this sense, white bottles with orange and green labels will be used.
  To mask the cinnamon smell of the capsule, the preparation in soft gelatin capsules with cinnamon oil will be used. This preparation, since the capsule is sealed, has no smell or flavor. For the placebo, soft gelatin capsules containing canola oil will be used.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Intervention (Experimental): 1000 mg orally of Cinnamomum Verum oil extract per day for 21-28 days
  Interventions: Drug: Cinnamomum Verum oil extract
- Placebo (Placebo Comparator): 400 mg orally of canola oil per day for 21-28 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cinnamomum Verum oil extract — one capsule of 1000 mg orally of Cinnamomum Verum oil extract per day for 21-28 days
  Other Names: cinnamon oil
  Arms: Intervention
Drug: Placebo — 400 mg PO Canola oil soft gel capsule
  Other Names: Canola oil; Kitchen oil
  Arms: Placebo

SUMMARY:
The purpose of the research protocol is to evaluate the effectiveness of Cinnamomum verum extract for the initiation of labor. Cinnamaldehyde ((E)-3-Phenylprop-2-enal) is an α, β unsaturated aromatic aldehyde, derived from cinnamon (Cinnamomum Verum oil) used as a flavoring; It is a clear yellowish liquid substance, with a strong odor and flavor. It is the main component of cinnamon (63%), giving it its physicochemical properties. Cinnamon has been an element of empirical use for the beginning of labor, however, its effectiveness has not been demonstrated.

Cinnamon has been reported for its ethnopharmacological properties in pregnancy, being used to facilitate childbirth, as a lactagogue and for postpartum recovery. In Honduras, its use has been reported to relieve nausea and vomiting during pregnancy, to reduce abdominal pain. , reduction of lower limb edema, to relieve anxiety during labor, as well as a lactagogue without convergent opinions.

DETAILED DESCRIPTION:
clinical trial of parallel groups of effectiveness, 2 groups will be taken, the intervention group will be administered capsules of Cinnamomum verum concentrate (1000 mg orally per day, a single dose) containing 67% cinnamaldehyde, one capsule per day will be administered (oral dose cinnamaldehyde lethal dose (LD50) of 1.15 g/kg), each capsule contains 1000 mg of Cinnamomum verum bark concentrate in soft gelatin capsules which are odorless and tasteless.

The control group will be administered canola oil capsules, a dose of 400 mg orally per day, a single dose per day. These soft gelatin capsules are odorless and tasteless.

Both capsules have identical physical characteristics. (they are soft gelatin capsules with the same color and smell)

ELIGIBILITY:
Inclusion Criteria:

1. Delivery of an informed consent form signed and dated by parents or guardian and patient
2. Declared willingness to comply with all study procedures and availability for the duration of the study.
3. provision of appropriate consent and assent
4. Willingness and ability to participate in study procedures
5. Patients under 18 years of age
6. Full-term pregnancies (37-41 Weeks of Gestation).
7. Nulliparity
8. Have your own cell phone
9. Know how to read and write
10. Residing in Tegucigalpa
11. Be in good general health, as evidenced by your medical history
12. Ultrasound with amniotic fluid index > 5 cm
13. Non Stress Test Reactive
14. Ability to take oral medication and be willing to comply with the cinnamon capsule regimen

Exclusion Criteria:

1. Current use of antihypertensive or hypoglycemic medications
2. Presence of non-curable chronic diseases prior to pregnancy or during pregnancy such as hypertension, diabetes, hypothyroidism
3. Premature rupture of membranes
4. Infections (urinary tract infection, chorioamnionitis) present at the time of the study (diagnosed with symptoms or leukocytes >12,500 or pathological urine examination)
5. Allergies to cinnamaldehyde or cinnamon, canola oil
6. Multiple pregnancy
7. Major fetal malformations
8. Fetal death
9. Non-cephalic presentation
10. Severe oligohydramnios (amniotic fluid index < 2 cm)
11. Having consumed or being consuming cinnamon products 7 days before the start of the study
12. Febrile illness within 7 days before starting to take cinnamon
13. Treatment with another investigational drug or other intervention within 7 days prior to the start of the intervention
14. Current smoker or tobacco use

Ages: 14 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Pregnancy
Enrollment: 70 (Estimated)
Dates: Start 2023-12-04 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Onset of labor | 21-28 days
  change in the time of onset of physiological phase 3 of the uterus (onset of labor)

SECONDARY OUTCOMES:
duration on labor | 24 hours
  change in duration of labor
cesarean section and/or instrumental delivery | 1-2 hours
  change in the rate of cesarean section and/or instrumental delivery
Neonatal complications | 28 days
  change of neonatal complications (apgar less than 7 at 5 minutes, meconium aspiration syndrome)
macrosomia | 1 hour
  change in incidence of macrosomia

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo A. Gutierrez Ramirez, MD, MSc, Principal Investigator — Universidad Nacional Autonoma de Honduras
Locations (1):
- Hospital Escuela, Tegucigalpa, Francisco Morazán Department, Honduras

IPD SHARING:
Plan to Share IPD: Yes
all the results
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: 1 year
Access Criteria: web data base